CLINICAL TRIAL: NCT04413188
Title: Effect of Warm Foot Bath on Their Sleep Quality and Comfort Level in Elderly Individuals: A Randomized-controlled Trial
Brief Title: A Warm Foot Bath, Sleep Quality and Comfort Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Hanife DURGUN, Principal Investigator, Ordu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HanifeB
Record Dates: First submitted 2020-05-27; First posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-06

CONDITIONS: Older People; Sleep Problems
MeSH Terms: conditions — Parasomnias

STUDY DESIGN:
Intervention Model Description: randomized controlled trail
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A warm foot bath group (Experimental): 65years, relative independent in daily life activities and literate, having a PSQI score of 5 or more and no communication problems.
  Interventions: Other: Warm foot bath
- Control group (No Intervention): 65years, relative independent in daily life activities and literate, having a PSQI score of 5 or more and no communication problems.

INTERVENTIONS:
Other: Warm foot bath — The participants in experimental group were asked to soak their feet in warm water (38-40°C) for 20 minutes one hour before their bedtimes for six weeks. A special foot bath (Beurer FB50 luxury foot bath spa with water heater) was used for this purpose. The bath is 10 cm deep; it keeps water at a constant temperature of 35-48°C for 15-60 minutes, has a display screen for water temperature and duration of use, and turns off automatically.
  Arms: A warm foot bath group

SUMMARY:
Objectives: To determine the effectiveness of a warm foot bath on sleep quality and comfort level among elderly individuals with sleep problems.

Design and methods: This study was a randomized controlled trial. A total of 217 elderly individual who stayed in two nursing homes. The sample consisted of 60 elderly individuals with sleep problem who were randomly assigned to either the warm foot bath group (n= 30) and control group (n=30).The study was completed with 60 elderly individuals. The primary outcome was an information questionnaire, the Pittsburgh Sleep Quality Index, the General Comfort Questionnaire and the Numerical Rating Scale.

DETAILED DESCRIPTION:
The age pyramid of the world population is changing, and as it does so, the percentage of elderly people is rapidly increasing. As one advances in age, it has been found that they tend to sleep latency later, have reduced time spent within crucial rapid eye movement (REM) sleep, and have reduced total duration and quality of sleep and sleep-related problems start to occur. The National Sleep Foundation The national sleep federation recommends 7-8 hours of sleep per day for the elderly. However, many elderly report that they sleep less than recommended and have difficulty sleep latency.

Sleeping is a significant action that affects individuals' daily lives as well as their quality of life. Sleep is required to meet the basic needs of daily life and comprises physiological, psychological, environmental and sociocultural dimensions. Sleep quality, which has been considered as increasingly significant in recent years, can be defined as feeling physically-fit, refreshed, and ready for a new day when waking up. Sleep quality consists of several quantitative aspects and measurements of sleep itself, such as the duration before sleep latency, the duration of sleep, the number of times a person wakes up in the night, as well as more subjective aspects such as the depth of sleep and the relaxing characteristic of sleep.

Such sleep-related problems may negatively affect an individual's comfort. Comfort is a basic need that comprises one of the cornerstones of holistic nursing care practice. Accordingly, solving sleep-related problems, increasing sleep quality, and ensuring comfort for the individuals concerned will require comprehensive nursing care. Pharmacological methods are the most commonly used approach in trying to resolve sleep-related problems. However, these methods have been insufficient as they do not provide a complete solution for sleep-related problems. Additionally, the side effects of these methods, which are obligatory for the affected individuals, are numerous, and this has paved the way for the development of non-pharmacological treatment methods. Relevant literature indicates methods such as eye masks, music therapy, massages, alternative and supplementary therapies, aromatherapy, and warm foot bath have all been successfully used to solve sleep-related problems among elderly people, thereby boosting their sleep quality and comfort.

Warm foot bath causes peripheral vasodilation and decreases core body temperatures. A negative relationship was found between core body temperature and inclination to sleep. Individuals' sleep latency decreases when body core temperature decreases thus, individuals' sleep quality and comfort level are increased. Warm foot bath as a non-pharmacological methods is a more practical and less expensive approach when compared with others.

The relevant literature demonstrated that the number of studies examining sleep quality and comfort among elderly people was limited. The literature included some studies that examined the use of relaxation exercises, back-massage practices, aromatherapy, and music therapy to improve sleep quality and comfort. However, the number of studies examining the effect of warm foot bath on sleep quality was found to be limited . The purpose of the trial was to investigate the effect of a warm foot bath on sleep quality and comfort level among elderly individuals with sleep problems. Our primary hypothesis was that the sleep quality of the intervention group would be better after 6 weeks than the control group. The secondary hypotheses were that the comfort levels of the intervention group would be better after 6 weeks than the control group

ELIGIBILITY:
Inclusion Criteria:

* 65 years and up
* relative independent in daily life activities
* literate
* having a PSQI score of 5 or more
* no communication problems.

Exclusion Criteria:

* who used sleeping drugs or diuretic drugs
* had peripheral artery diseases
* neurological diseases.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Sleep quality: Pittsburgh Sleep Quality Index (PSQI) | before applying the first foot bath
  The Pittsburgh Sleep Quality Index (PSQI) This index was developed by Buysse and colleagues to evaluate individuals' sleep quality and sleeping disorders over a month. The scale consists of 24 items, 19 of these items are related to self-reporting and are answered by the respondents. This is composed of 19 questions which reflect seven major components. The last five items of the index (11a, 11b, 11c, 11d, and 11e) are answered by the partners or roommates of the participants, and these items are not included in the scoring. Each item is scored with points ranging from 0 to 3, with 0 indicating a "good" score and 3 indicating a "poor" score. Accordingly, higher total scores indicate poor sleep quality; scores of 0-4 indicate good sleep quality, and scores of 5-21 suggest poor sleep quality
Sleep quality: Pittsburgh Sleep Quality Index (PSQI) | six weeks after the first foot bath
  The Pittsburgh Sleep Quality Index (PSQI) This index was developed by Buysse and colleagues to evaluate individuals' sleep quality and sleeping disorders over a month. The scale consists of 24 items, 19 of these items are related to self-reporting and are answered by the respondents. This is composed of 19 questions which reflect seven major components. The last five items of the index (11a, 11b, 11c, 11d, and 11e) are answered by the partners or roommates of the participants, and these items are not included in the scoring. Each item is scored with points ranging from 0 to 3, with 0 indicating a "good" score and 3 indicating a "poor" score. Accordingly, higher total scores indicate poor sleep quality; scores of 0-4 indicate good sleep quality, and scores of 5-21 suggest poor sleep quality
Comfort level | six weeks after the first foot bath
  The General Comfort Questionnaire (GCQ) This questionnaire was developed by Katharine Kolcaba in 1992 to determine individuals' comfort needs and evaluate nursing interventions that might be employed to ensure and increase such comfort. The GCQ uses a four-point Likert type scale and consists of 48 items. The lowest score that can be obtained from the scale is 48, the highest score is 192. The total score obtained from the scale was divided by 48 (the number of the items in the scale) to determine the score's mean value which was presented as a score between one and four. The GCQ was adapted for use in a Turkish context by Kuguoğlu and Karabacak in 2004. The Cronbach's alpha coefficient of the original scale was 0.88; in the study by Kuguoglu and Karabacak, it was 0.85. The present study derived a Cronbach's alpha coefficient of 0.68 prior to experimental and 0.75 after experimental.
Dailiy sleep quality: The Numerical Rating Scale (NRS) | Daily for six weeks
  The Numerical Rating Scale (NRS) This scale was prepared as a form incorporating a scale; it was then used by individuals who were able to mark and assess their personal sleep quality each day. The NRS asks patients to choose the number from 0 to 10 that best represents their sleep with 0 representing a poor night's sleep, and 10 representing a good night's sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Hanife Durgun, Dr, Principal Investigator — Ordu State Hospital

IPD SHARING:
Plan to Share IPD: No